CLINICAL TRIAL: NCT02986035
Title: Effectiveness of ECA Cream on Calcifying Shoulder Tendinitis
Acronym: ECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Collaborators: PRODUCTOS SANITARIOS ECA-RVB SLI (Unknown)
Responsible Party: Principal Investigator, Lluís Guirao, PhD, Consorci Sanitari del Maresme
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46/16
Record Dates: First submitted 2016-11-28; First posted 2016-12-07 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Calcifying Shoulder Tendinitis
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Other: ECA cream

INTERVENTIONS:
Other: ECA cream

SUMMARY:
This pilot trail aims to assess the effectiveness of ECA cream in the treatment of calcifying shoulder tendinitis in terms of:

1. Reduction or removal of shoulder calcifications
2. Functional improvements
3. Pain improvements 10 subjects will be assessed prior and 1 and 2 months post intervention onset. The intervention will consist in the application of the ECA cream in the affected shoulder twice a day during 1 month.

ELIGIBILITY:
Inclusion Criteria:

* patients >=18 years
* diagnosed of calcifying shoulder tendinitis diagnosed by a medical specialist (rehabilitation, orthopedic surgeon or rheumatologist) by x-ray
* with disease evolution of more than 3 months and less than 12 months
* that give their informed consent by writing

Exclusion Criteria:

* Previous shoulder surgery patients
* Patients with shoulder affections treated with shockwaves or corticosteroid injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Presence of shoulder calcifications | 2 months
  X-ray
Size of shoulder calcifications | 2 months
  Ultrasonography

SECONDARY OUTCOMES:
Shoulder functionality | 1 and 2 months
  Constant Scale
Shoulder pain | 1 and 2 months
  Pain VAS (Visual Analogue Scale )

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari del Maresme, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No